CLINICAL TRIAL: NCT00958737
Title: A Phase III Randomized Trial Investigating the Duration of Adjuvant Therapy(3 Versus 6 Months) With the Modified FOLFOX 6 or XELOX Regimens for Patients With Stage III Colon Cancer
Brief Title: Combination Chemotherapy for 3 Months or 6 Months in Treating Patients With Stage III Colon Cancer
Acronym: IDEA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEA-C09-1; 2009-010384-16 (EudraCT Number); EU-20957 (Other: EU Clinical Trials Register)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Folfox protocol; Leucovorin; Oxaliplatin; Capecitabine; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive modified FOLFOX 6 comprising oxaliplatin IV 85 mg/m² over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1. Treatment repeats every 14 days for 6 courses (3 months).
  Patients receive CAPOX comprising oxaliplatin IV 130 mg/m² over 2 hours (day 1 every 3 weeks) in combination with capecitabine, which will be administered orally at a dose of 1000 mg/m2 twice-daily (equivalent to a total daily dose of 2000 mg/m2), with first dose the evening of day 1 and last dose the morning of day 15, given as intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment)
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX
- Arm II (Experimental): Patients receive modified FOLFOX 6 or CAPOX as in arm I. Treatment repeats every 14 days for 12 courses (6 months)or regarding CAPOX every 21 days for 8 courses (6 month).
  Interventions: Drug: FOLFOX regimen; Drug: CAPOX

INTERVENTIONS:
Drug: FOLFOX regimen — 6 or 12 treatments of FOLFOX (FOLFOX4 or modified FOLFOX6 (mFOLFOX6))
  Other Names: folinic acid, infusional fluorouracil, and oxaliplatin
Drug: CAPOX — 4 or 8 cycles
  Other Names: capecitabine plus oxaliplatin; XELOX

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving more than one drug (combination chemotherapy) is more effective when given for 3 months or 6 months in treating patients with colon cancer.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy for 3 months to see how well it works compared with giving combination chemotherapy for 6 months in treating patients with stage III colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective

* To assess whether a 3-month modified FOLFOX 6 or XELOX treatment is not inferior to a 6-month modified FOLFOX 6 or XELOX treatment in terms of disease free survival (DFS) in patients with radically resected stage III colon cancer.

Secondary Objectives

* To assess whether 3-month modified FOLFOX 6 (6 cycles) or XELOX (4 cycles) treatment is not inferior to 6-month modified FOLFOX 6 (12 cycles) or XELOX (8 cycles) treatment in terms of overall survival (OS) in patients with radically resected stage III colon cancer
* To evaluate the safety profiles of the treatment groups

Tertiary Objectives

* For patients who signed a specific informed consent, blood and tumour tissue samples will be stored, registered, and centralized in a data bank for translational research projects that will be further determined according to the literature and scientific knowledge at the time of the end of inclusion. (exploratory)
* An economic evaluation at the country level will be conducted alongside the clinical evaluation. (exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to center, T stage (1 or 2 vs 3 vs 4), N stage (1 vs 2), performance status (0 vs 1 vs 2), and age (< 70 years vs ≥ 70 years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive modified FOLFOX 6 comprising oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1. Treatment repeats every 14 days for 6 courses (3 months).
* Arm II: Patients receive modified FOLFOX 6 as in arm I. Treatment repeats every 14 days for 12 courses (6 months).

Blood and tumor samples may be collected at baseline for pharmacogenetic and other analyses.

After completion of study treatment, patients are followed up every 6 months for 8 years.

ELIGIBILITY:
Inclusion criteria:

* Patients who have undergone surgery for colon cancer, defined as a tumor location >12 cm from the anal verge by endoscopy and/or above the peritoneal reflection at surgery (high rectum), without gross or microscopic evidence of residual disease after surgery with curative intent.
* Histologically confirmed AJCC/UICC stage III adenocarcinoma colon cancer.
* Age >18 years.
* Curative surgery and no more than 8 weeks prior to randomization.
* ECOG performance Status (ECOG-PS) <2.
* Signed written informed consent obtained prior to any study specific procedures.
* CEA ≤ 10 ng/ml (2 X normal value).
* Post-menopausal women or women willing to accept the use of an effective contraceptive regimen during the treatment period and up to 1 month after the end of the study treatment. All non postmenopausal women should have a negative pregnancy test within 72 hours prior to randomization. Men should accept to use an effective contraception during the treatment period, and up to 1 month after the end of the study treatment.
* Registration in a national health care system (CMU included).

Exclusion criteria:

Macroscopic or microscopic evidence of residual tumor (R1 or R2 resections). Patients should never have had any evidence of metastatic disease (including presence of tumor cells in ascites or peritoneal carcinomatosis resected "en bloc").

* Cancer of low or medium rectum with tumor location < 12 cm from the anal verge by endoscopy.
* Other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix).
* Pregnant or lactating women
* Clinically relevant cardiovascular disease (for example: ischemic myocardial infarction in the last year and/or unstable ischemic cardiopathy).
* History or current evidence on physical examination of central nervous system disease or peripheral neuropathy ≥ grade 1 Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0.
* Known hypersensitivity reaction to any of the components of study treatments.
* Current or recent (within 28 days prior to randomization) treatment with another investigational drug.
* Subject unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-05-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years after randomisation
  DFS, defined as the time from random assignment to relapse or death, whichever occurred first. Secondary colorectal cancers were regarded as DFS events, whereas noncolorectal cancers were disregarded in the analysis.

SECONDARY OUTCOMES:
Overall survival (OS) | Death from randomization; up to 7 years after randomization
  The time from the date of randomization to the date of death from any cause
Safety profile | Assessed up to 6 months after randomisation
  All grade and severe toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Treatment compliance | Until 3 months or 6 months (according randomization arm)
  duration, dose intensity, and dose in mg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Andre, MD, Principal Investigator — GERCOR - Multidisciplinary Oncology Cooperative Group
Locations (1):
- GERCOR Groupe Cooperateur Multidisciplinaire en Oncologie, Paris, France

REFERENCES:
- [Result] Andre T, Vernerey D, Mineur L, Bennouna J, Desrame J, Faroux R, Fratte S, Hug de Larauze M, Paget-Bailly S, Chibaudel B, Bez J, Dauba J, Louvet C, Lepere C, Dupuis O, Becouarn Y, Mabro M, Egreteau J, Bouche O, Deplanque G, Ychou M, Galais MP, Ghiringhelli F, Dourthe LM, Bachet JB, Khalil A, Bonnetain F, de Gramont A, Taieb J; for PRODIGE investigators, GERCOR, Federation Francaise de Cancerologie Digestive, and UNICANCER. Three Versus 6 Months of Oxaliplatin-Based Adjuvant Chemotherapy for Patients With Stage III Colon Cancer: Disease-Free Survival Results From a Randomized, Open-Label, International Duration Evaluation of Adjuvant (IDEA) France, Phase III Trial. J Clin Oncol. 2018 May 20;36(15):1469-1477. doi: 10.1200/JCO.2017.76.0355. Epub 2018 Apr 5. PMID 29620995
- [Derived] Taieb J, Souglakos J, Boukovinas I, Falcoz A, Pages F, Messaritakis I, Bennouna J, Artru P, Louvet C, Lepere C, Emile JF, Bouche O, Mazard T, Vernerey D, Vogiatzoglou K, Tzardi M, Sharma S, Liu MC, Sethi H, Andre T, Galon J, Laurent-Puig P. Combined Analyses of Circulating Tumor DNA and Immunoscore in Patients With Stage III Colon Cancer: A Post Hoc Analysis of the PRODIGE-GERCOR IDEA-France/HORG-IDEA-Greece Trials. J Clin Oncol. 2025 May;43(13):1564-1577. doi: 10.1200/JCO.24.00648. Epub 2025 Feb 4. PMID 39903903
- [Derived] Gallois C, Sroussi M, Andre T, Mouillet-Richard S, Agueeff N, Mulot C, Vernerey D, Louvet C, Bachet JB, Dourthe LM, Mazard T, Jary M, Coutzac C, Lecaille C, Tabernero J, Van Laethem JL, Lepage C, Emile JF, de Reynies A, Taieb J, Laurent-Puig P. Prognostic Models From Transcriptomic Signatures of the Tumor Microenvironment and Cell Cycle in Stage III Colon Cancer From PETACC-8 and IDEA-France Trials. J Clin Oncol. 2025 May 20;43(15):1765-1776. doi: 10.1200/JCO.23.02262. Epub 2025 Jan 31. PMID 39889251
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Delattre JF, Cohen R, Henriques J, Falcoz A, Emile JF, Fratte S, Chibaudel B, Dauba J, Dupuis O, Becouarn Y, Bibeau F, Taieb J, Louvet C, Vernerey D, Andre T, Svrcek M. Prognostic Value of Tumor Deposits for Disease-Free Survival in Patients With Stage III Colon Cancer: A Post Hoc Analysis of the IDEA France Phase III Trial (PRODIGE-GERCOR). J Clin Oncol. 2020 May 20;38(15):1702-1710. doi: 10.1200/JCO.19.01960. Epub 2020 Mar 13. PMID 32167864
- See also: IDEA France phase III trial — https://pubmed.ncbi.nlm.nih.gov/29620995/